CLINICAL TRIAL: NCT05759923
Title: An Open-label, Multicentre, Dose-escalation, First-in-human Phase I Study to Evaluate Safety, Tolerability and Antineoplastic Activity of OATD-02 in Patients with Selected Advanced And/or Metastatic Solid Tumours (colorectal Cancer, Ovarian Cancer, Pancreatic Cancer or Renal Cell Carcinoma)
Brief Title: First-in-human Phase I Study to Evaluate Safety, Tolerability and Antineoplastic Activity of OATD-02 in Patients with Selected Advanced And/or Metastatic Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Molecure S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OATD-02-C-01
Record Dates: First submitted 2023-02-09; First posted 2023-03-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-07

CONDITIONS: Advanced Ovarian Carcinoma; Advanced Renal Cell Carcinoma; Advanced Pancreatic Carcinoma; Advanced Colorectal Carcinoma; Metastatic Pancreatic Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Ovarian Carcinoma
Keywords: solid tumors; renal cancer; ovarian cancer; pancreatic cancer; colorectal cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Renal Cell; Ovarian Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OATD-02 (Experimental)
  Interventions: Drug: OATD-02

INTERVENTIONS:
Drug: OATD-02 — Boin Design Scheme will be applied for dose escalation. Dose will start with 2.5mg o.d., the desicion about dose escalations will be made based on the occurence of DLT

SUMMARY:
The goal of this clinical trial is to learn if the OATD-02 administration (orally) in monotherapy is safe and has the pharmacodynamic potential to restore and enhance tumour responses to immunotherapy through increased arginine levels or intrinsic anti-tumour activity in participants with advanced metastatic colorectal cancer, ovarian cancer, renal cancer or pancreatic cancer.

DETAILED DESCRIPTION:
In this study, subjects suitable for enrollment will be identified by the investigators involved in the study. These subjects will be identified through contact with these investigators and referred for enrollment per protocol. This protocol will include determining enrollment suitability based on inclusion and exclusion criteria.

Study scheme is based on Modified Bayesian Optimal Interval (BOIN) design.

The BOIN design works by partitioning the probability of toxicity into a set of intervals. This design makes dose-selection decisions determined by the interval in which the probability of toxicity for the current dose is believed to reside. BOIN seeks a dose with probability of toxicity close to some pre-specified target level.

Total number of patients will be 30 (plus 10 replacements if Dose Limiting Toxicity (DLT) is not evaluable).

Study treatment will be up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and complying with protocol requirements.
2. Male or female patient aged ≥18 years at Screening.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Histologically or cytologically confirmed advanced and/or metastatic colorectal cancer, renal cell cancer, or pancreatic cancer or recurrent serous ovarian cancer (platinum-resistant/ineligible to receive platinum-based chemotherapy), that either progressed or relapsed after all relevant standard of care cancer therapies (at least 1 line of systemic cancer therapy).
5. Written informed consent given by the patient before the initiation of any study procedures.

Exclusion Criteria:

1. Unable to take oral medications.
2. Clinically active central nervous system metastases and/or carcinomatous meningitis.
3. Major surgery within 30 days before the first IMP dose.
4. Pregnant or breastfeeding women.
5. Known allergy to excipients of the IMP.
6. Severe, uncontrolled systemic disease which in the opinion of the investigator, would compromise the safety of the patient or the patient's ability to participate in the study.
7. Participation in another clinical study within 4 weeks before the first IMP dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Nature, frequency and severity of adverse events (AEs) | 6 months
Occurence of DLTs | 6 months

SECONDARY OUTCOMES:
PK parameters for OATD-02: CMax | 6 months
Anti-tumour activity parameters (Objective Response Rate (ORR), Duration of Response (DoR), PFS (Progression Free Survival) followed up to the End of Study Visit | 6 months
PK parameter: Tmax | 6 months
PK parameter Cmin | 6 months
PK parameter: AUCO-24 | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Site, Otwock, Masovian Voivodeship
  - SIte, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: No